CLINICAL TRIAL: NCT02155452
Title: Understanding the Mechanisms of ALA-induced Fluorescence in Malignant Gliomas - Exploring the Biological Basis of Tumoral Heterogeneity.
Brief Title: Fluorescence and Glioma Heterogeneity
Acronym: ALAglioma
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Aliasgar V Moiyadi, Prof Neurosurgery, Tata Memorial Hospital
Other Study IDs: TMC- ACTREC IRB project no 139
Record Dates: First submitted 2014-05-17; First posted 2014-06-04 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Malignant Gliomas
Keywords: ALA; Malignant gliomas
MeSH Terms: conditions — Glioma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The heterogeneity of fluorescence within malignant gliomas by sampling tissues from these variable areas within the same tumor. These tissue samples will then be subjected to pathological and biological analysis to assess proteins related to ALA metabolism and correlated with the fluorescence emitted as well as levels of protoporphyrin IX in the tissues.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- With ALA: Patients with malignant glioma. 25 patients will be provided the ALA for inducing fluorescence
  Interventions: Procedure: ALA
- Without ALA: 5 tumor tissue samples from ACTREC tumor tissue repository will be obtained. These would be malignant gliomas or other brain tumor samples where ALA is usually not administered and will be used as controls and for calibration purposes

INTERVENTIONS:
Procedure: ALA — Prior to surgery all patients would receive freshly prepared solution of 5-ALA, 20 mg/kg bodyweight dissolved in 100 ml of potable water orally approximately 4 hours (range 4-6 hrs) before the commencement of anesthesia induction for surgery.
  The surgery would then be performed with the help of navigation. After craniotomy, the navigation software would be used to identify the selected target areas based on the preoperative images (MR as well as PET when available) and directed image-guided biopsies from these representative areas will be collected for histological evaluation
  Other Names: 5- ALA
  Groups: With ALA

SUMMARY:
The investigators aim to study the heterogeneity of fluorescence within malignant gliomas by sampling tissues from these variable areas within the same tumor. These tissue samples will then be subjected to pathological and biological analysis to assess proteins related to ALA metabolism and correlated with the fluorescence emitted as well as levels of protoporphyrin IX in the tissues.

DETAILED DESCRIPTION:
Malignant gliomas are the commonest malignant brain tumors but are extremely challenging to treat. Neuro-oncology has seen little progress in its treatment despite extensive research. Extent of resection remains a very important prognostic factor in these tumors. Better the resection, better the outcomes. However resecting these tumors is not very easy primarily due to their infiltrative nature and difficulty in discerning tumor boundaries intraoperatively. Fluorescence guided resection (FGR) has recently been shown to be a very important and useful adjunct in maximizing this goal. FGR involves administration of aminolevulinic acid (ALA) to the patient prior to surgery. The ALA is converted to protoporphyrin IX (PPIX) in glioma cells. The PPIX is a fluorophore and can be visualized intraoperatively using a suitably modified microscope. Neurosurgeons can then resect the tumor radically guided by this fluorescence which is superior to the conventional microscopic resection. Selective PPIX accumulation in glioma cells is the key to the accuracy of this technique. The biological basis of selectivity of PPIX accumulation within glioma cells is however poorly understood. Various mechanisms could be involved starting from variable transport (related to blood-brain barrier properties), differential uptake (governed by active transport mechanisms) and differential metabolism within the cell. Understanding these mechanisms can lead to refinements in this strategy, overcoming its present limitations and development of methods to extend its scope.

ELIGIBILITY:
Inclusion Criteria:

Per-primum glioma

* Adults (18-65 years)
* Radiologically suspected malignant gliomas
* Variable contrast enhancement on MRI (patchy and/or non-uniform)
* Eligible for surgical therapy (craniotomy NOT stereotactic biopsy )
* No contraindication for surgery

Exclusion Criteria:

* Poor general condition (KPS < 70)
* Prior treatment (except biopsy)
* Compromised renal/hepatic function
* Immunocompromised status
* Known photosensitivity / allergy to 5-ALA

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignant glioma
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Degree of fluorescence | At the time of surgery within 72 hours
  1. Degree of fluorescence in different tumor regions
  2. PPIX Qualification

SECONDARY OUTCOMES:
High throughput proteomic screening of tissue samples | Postoperatively within 1 week of the excision
  -A quantitative approach will be undertaken to compare the proteome profile

CONTACTS AND LOCATIONS:
Overall Officials: Aliasgar V Moiyadi, MCh DNB, Principal Investigator — neurosurgeon
Locations (1):
- Advanced Centre for Treatment, Research & Education in Cancer (ACTREC), Navi Mumbai, Maharashtra, India